CLINICAL TRIAL: NCT04659447
Title: Clinical Study of Platelet-rich Plasma Promoting Tendon-bone Healing in Anterior Cruciate Ligament Reconstruction
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Beijing Tsinghua Chang Gung Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12017B3003
Record Dates: First submitted 2020-11-23; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Sports Injury
Keywords: Anterior Cruciate Ligament Tear; platelet-rich plasma
MeSH Terms: conditions — Athletic Injuries; Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet-Rich Plasma (Experimental): Four semitendinosus tendons and gracilis tendons are prepared. 4 ml platelet-rich plasma is completely absorbed by a gelatin sponge and fixed in the center of the four tendons. 4-0 absorbable line is used for fixation.Then we use conventional surgical techniques to reconstruct the ACL.
  Interventions: Drug: Platelet-Rich Plasma
- control group (No Intervention): We performed conventional surgical techniques to reconstruction without using platelet-rich plasma.

INTERVENTIONS:
Drug: Platelet-Rich Plasma — 36 ml of peripheral blood is extracted from patients, and 4 ml of 3.8% sodium citrate is added for anticoagulation. After centrifugation for 2 times, 4 ml platelet-rich plasma will be prepared.Four semitendinosus tendons and gracilis tendons are prepared.
  Arms: Platelet-Rich Plasma

SUMMARY:
Anterior cruciate ligament (ACL) injury is a common knee injury, which seriously affects the living ability and sport level of the injured. ACL reconstruction is the main method to treat ACL injury. Due to the reconstructive ligament needs a tendon bone healing and ligament maturation, therefore, in the ACL anatomical study, reconstruction surgery and reconstruction materials under the condition of constant progress, how to improve the ACL reconstruction of tendon bone healing and shorten the time of the ligament mature, improve the clinical effect of ACL reconstruction, has become the focus in the ACL reconstruction.

Autologous platelet-rich plasma (PRP) is full of growth factors and bioactive factors, which has the function of promoting tissue healing, anti-inflammatory and analgesic effects. At the same time of anterior cruciate ligament reconstruction, using autologous PRP in the bone channel might promote tendon bone healing and ligament maturing after ACL reconstruction, promote the recovery of proprioception, prevent bone channel expanding, shorten the postoperative recovery time, speed up the patients recovery exercise ability, improve the clinical effect of ACL reconstruction.

In this study, patients with ACL injuries were randomly divided into two groups: one group underwent ACL anatomical reconstruction, and the other group underwent ACL anatomical reconstruction with PRP. Various clinical scores, KT-2000, Biodex and imaging tests were used to evaluate the differences in the clinical effects of the two surgical methods in terms of postoperative pain, joint swelling, knee function, joint stability, muscle strength recovery, bone channel expanding, ligament vasinization, and ligament maturation.

ELIGIBILITY:
Inclusion Criteria:

* History of knee injury
* History of knee instability
* Anterior drawer test (+), or / and Lachman test (+)
* The tear of anterior cruciate ligament was confirmed by MRI

Exclusion Criteria:

* The injury of other ligaments of knee joint, such as complex posterior cruciate ligament injury, lateral collateral ligament injury and medial collateral ligament injury above III degree
* Patients with meniscus removed
* Patients with moderate to severe articular cartilage injury
* Patients with complex nerves and blood vessels injury
* Patients with compound intra - and periarticular fractures of the knee
* Patients with intra or periarticular fractures of the knee
* Patients with contralateral knee instability
* Patients with severe cardiovascular and cerebrovascular diseases

Ages: 15 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2021-11-09 (Estimated); Study Completion 2021-11-09 (Estimated)

PRIMARY OUTCOMES:
tendon bone healing and ligament maturing | CT and MRI were performed on the fourth day after operation
  The diameter of bone canal was evaluated by CT, it is measured in millimeters (mm).
  The tendon bone healing and ligament maturing was evaluated by MRI. According to the same level of anterior cruciate ligament, femoral canal, posterior cruciate ligament, background noise, with the diameter of 3.3 mm as the center, the lowest signal value point was measured, and the final point was compared to obtain the Signal-Noise Ratio.
tendon bone healing and ligament maturing | CT and MRI were performed on one year after operation
  The diameter of bone canal was evaluated by CT, it is measured in millimeters (mm).
  The tendon bone healing and ligament maturing was evaluated by MRI. According to the same level of anterior cruciate ligament, femoral canal, posterior cruciate ligament, background noise, with the diameter of 3.3 mm as the center, the lowest signal value point was measured, and the final point was compared to obtain the Signal-Noise Ratio.
proprioception and Knee joint function | 3 months after the operation
  KT-2000, it was used to assess the stability of the tibia and the results were expressed in millimeters.
  Biodex, it is used to assess the strength and function of joints. The contralateral knee joint was taken as the reference. The percentage of strength between the affected knee joint and the contralateral knee joint was obtained
proprioception and Knee joint function | 6 months after the operation
  KT-2000, it was used to assess the stability of the tibia and the results were expressed in millimeters.
  Biodex, it is used to assess the strength and function of joints. The contralateral knee joint was taken as the reference. The percentage of strength between the affected knee joint and the contralateral knee joint was obtained
proprioception and Knee joint function | 1 year after the operation
  KT-2000, it was used to assess the stability of the tibia and the results were expressed in millimeters.
  Biodex, it is used to assess the strength and function of joints. The contralateral knee joint was taken as the reference. The percentage of strength between the affected knee joint and the contralateral knee joint was obtained
Knee pain | 3 months after the operation
  Visual Analog Score for pain, it is used to assess the patient's pain, the full score is 10.
Knee pain | 6 months after the operation
  Visual Analog Score for pain, it is used to assess the patient's pain, the full score is 10.
Knee pain | 1 year after the operation
  Visual Analog Score for pain, it is used to assess the patient's pain, the full score is 10.

REFERENCES:
- [Derived] Gong H, Huang B, Zheng Z, Fu L, Chen L. Clinical Use of Platelet-Rich Plasma to Promote Tendon-Bone Healing and Graft Maturation in Anterior Cruciate Ligament Reconstruction-A Randomized Controlled Study. Indian J Orthop. 2022 Jan 27;56(5):805-811. doi: 10.1007/s43465-021-00533-z. eCollection 2022 May. PMID 35103026